CLINICAL TRIAL: NCT05947136
Title: PASCA-MM Study. Impact of the PASCA (PArcours de Santé au Cours du CAncer) Program on Complications Associated With Multiple Myeloma and/or Its Treatments in the Context of a First Hematopoietic Stem Cell Autograft, in Adults Aged 18 to 70.
Acronym: PASCA -MM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PASCA-MM (ET22000285)
Record Dates: First submitted 2023-07-07; First posted 2023-07-17 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Multiple Myeloma; Complication
Keywords: Multiple Myeloma; Complications; Detection; Intervention; Autologous stem cell transplant; Randomized controlled trials
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): For both the 7 complications of interest (primary objective) and the 13 secondary complications (secondary objective), specific and proactive referrals will be made systematically after each detection visit according to the level of risk, estimated on the basis of decision trees (management guide) and via the dedicated PASCA network of healthcare professionals, to initiate early treatment and follow-up where necessary.
  Interventions: Behavioral: Interpretation of the results from the detection visit; Behavioral: Explaining detection results and referrals to the patient; Behavioral: Early medical care through the network
- Control group (Active Comparator): For both the 7 complications of interest (primary objective) and the 13 secondary complications (secondary objective): all the data from each detection visit will be sent to the referring forwarded to the referring onco-haematologists, so that they can initiate their own management.
  Interventions: Behavioral: Transmission of results from each detection visit to the referring onco-haematologists - Control Group

INTERVENTIONS:
Behavioral: Interpretation of the results from the detection visit — - An interpretation of the results of the detection tests concerning
  * the 7 complications of interest assessed at T1, T2, T3 and T4 ;
  * the 13 secondary complications assessed at T1, T3 and T4. This interpretation will be based on decision trees (1 tree/complication) to guide investigators in their decision-making and to standardise orientations;
  Arms: Intervention group
Behavioral: Explaining detection results and referrals to the patient — Explanation of results and directions to the patient using plain language;The aims of this call are as follows:
  * Clearly explain the results of the detection visit and the action to be taken for each referral;
  * Evaluate the help to be given to the patient. This help will consist of making bookings with a healthcare professional in the PASCA network;
  * Reassure patients about their results, but also make them aware of the importance of taking action to improve or prevent the onset of complications.
  Arms: Intervention group
Behavioral: Early medical care through the network — Early, proactive medical care through a network of dedicated healthcare professionals.
  Arms: Intervention group
Behavioral: Transmission of results from each detection visit to the referring onco-haematologists - Control Group — For both the 7 complications of interest (primary objective) and the 13 secondary complications (secondary objective): all the data from each detection visit will be sent to the referring onco-haematologists, so that they can initiate their own management.
  Arms: Control group

SUMMARY:
This is a prospective, multicentre, phase III, randomised, controlled intervention study.

Two groups of patients with equal numbers will be studied and each patient will be allocated to one of the two groups described below by randomisation (ratio 1:1).

Each patient will be allocated to one of the two groups described below by randomisation (ratio 1:1).

- PASCA interventional group

For both the 7 complications of interest (primary objective) and the 13 secondary complications (secondary objective), a specific and proactive referral will be made systematically after each screening assessment, depending on the level of risk, estimated according to decision trees (management guide) and through the dedicated PASCA network of healthcare professionals, in order to initiate early treatment and follow-up if necessary.

- Control group

For the 7 complications of interest (primary objective) as well as for the 13 complications (secondary objective): all the data from each identification check-up will be sent to the onco-haematological transmitted to the referring onco-haematologists, so that they can initiate their own management.

=> For all patients, regardless of group

All patients will receive four screening assessments covering the 7 complications of interest and 13 secondary complications:

* Visit No.1 (T1), 1-2 months after the autologous haematopoietic stem cell transplantation (aHSCT), corresponding to the patient's visit to his or her Multiple Myeloma (MM) monitoring consultation and/or the start of his or her consolidation treatment.
* Visit No.2 (T2), 4 months after aHSCT, corresponding to a patient's visit for the end of consolidation treatment;
* Visit No.3 (T3), 14 months after the last aHSCT, corresponding to a visit by the patient during his or her maintenance treatment;
* Visit No.4 (T4), 24 months after the last aHSCT, corresponding to a visit by the patient for a MM monitoring consultation.

DETAILED DESCRIPTION:
After each screening visit, all patients randomised to the intervention group will receive the PASCA intervention:

1. An interpretation of the results of the screening tests concerning

   * the 7 complications of interest assessed at T1, T2, T3 and T4 ;
   * the 13 secondary complications assessed at T1, T3 and T4. This interpretation will be based on decision trees (1 tree/complication) to guide investigators in their decision-making and to standardise orientations;
2. Explanation of results and referrals to the patient using plain language, by a phone call, ;
3. Early, proactive care via a dedicated network of healthcare professionals.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old and ≤ 70 years old.
2. Patient treated in an investigation center.
3. Symptomatic multiple myeloma eligible for autologous hematopoietic stem cell transplantation (HSCT).
4. In stringent complete response, complete response, very good complete response, or partial before HSCT.
5. First induction-type treatment (Isa-KRD/dara-VRD/dara-VTD/VRD/VTD), intensification therapy with melphalan, HSCT, consolidation, maintenance including at least one drug immunomodulator.
6. ECOG performance status WHO ≤ 2.
7. No history or coexistence of other primary cancer apart from basal cell cancer cutaneous
8. Able to understand, read and write French.
9. Having signed and dated the informed consent.

Exclusion Criteria:

1. Unable to be monitored for medical, social, family, geographical or psychological, throughout the duration of the study.
2. Deprived of liberty by court or administrative decision.
3. Not affiliated with a health insurance plan.
4. Not having declared an attending physician.
5. Not domiciled in the Auvergne-Rhône-Alpes region or in the Saône-et-Loire department.
6. Not available and/or not willing to participate in the project for the entire duration of the study.
7. Pregnant women, breastfeeding women, people in emergency situations, people incapable of personally giving their consent including adults under guardianship

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2027-06-14 (Estimated); Study Completion 2027-09-14 (Estimated)

PRIMARY OUTCOMES:
change from Baseline high blood pressure | month 2, month 4, month 14 and month 24
  blood pressure ≥ 140/90 mmHg measured in the investigating center and persisting over time
Change from Baseline chronic kidney failure incidence at 24 months | month 2, month 4, month 14 and month 24
  diagnosed on the basis of 2 blood tests carried out within 3 months with the same technique showing either:
  * a decrease in GFR to < 60ml/min/1.73m2, estimated from serum creatinine using the CKD-EPI equation (Chronic Kidney Disease EPIdemiology collaboration, Levey, 2009),
  * positive proteinuria or albuminuria (albuminuria/creatinine ratio),
  * haematuria with a GR > 10/mm3 or 10,000/ml (after eliminating a urological cause),
  * leucocyturia with a WBC >10/mm3 or 10,000/ml (in the absence of infection),
  * a morphological abnormality on renal ultrasound: size asymmetry, bumpy contours, small kidneys or large polycystic kidneys, nephrocalcinosis, cyst.
  The evolutionary character corresponds to one of the following situations:
  * Annual decline in GFR ≥ 5 ml/min/1.73 m²/year: GFR year n - GFR year n+1
  * Presence of albuminuria,
  * Poorly controlled arterial hypertension
Change from Baseline chronic pain incidence at 60 months | month 2, month 4, month 14 and month 24
  pain felt for more than 3 months by the patient with an intensity on the Visual Analogue Scale (VAS) ≥ 3
Change from Baseline sexual disorders incidence at 24 months | month 2, month 4, month 14 and month 24
  at least one perceived problem among the following:
  * disorders of desire,
  * arousal/erection disorders in men,
  * arousal disorders (insufficiency) in women,
  * Orgasm disorders in women
Change from Baseline osteoporosis incidence at 24 months | month 2, month 14 and month 24
  T-score evaluated by osteodensitometry, on the lumbar spine and upper end of the femur
Change from Baseline chronic fatigue incidence at 24 months | month 2, month 4, month 14 and month 24
  Questionnaire "MFI-20" (Multidimensional Fatigue Inventory)
Change from Baseline severe anxiety disorder incidence at 24 months | month 2, month 4, month 14 and month 24
  Questionnaire "HADS-D" (Hospital Anxiety and Depression scale)

SECONDARY OUTCOMES:
Change from Baseline depressive events incidence at 24 months | month 2, month 4, month 14 and month 24
  Defined by at least two main depressive symptoms, associated with at least two symptoms additional information, according to the 2017 HAS recommendation "Characterized depressive episode in adults
  : care in first resort".
Change from Baseline physical deconditioning incidence at 24 months | month 2, month 14 and month 24
  Defined by at least two tests among the 6 min Walk Test (TDM6), Handgrip-test, 60s Sit-to-stand, Flamingo test, with usual values below the norms defined by their authors, according to age and sex
Change from Baseline cognitive problems incidence at 24 months | month 2, month 14 and month 24
  Positive score on at least one of the sub-dimensions of the Functional questionnaire Cancer Therapy Assessment - Cognitive Function (FACT-COG)
Change from Baseline hypogonadism incidence at 24 months | month 2, month 14 and month 24
  Presence of clinical signs as defined by the International Society for Sexual Medicine
  A value below the lower limit on at least one of the following blood assay:
  * level of total testosterone
  * level of bioavailable testosterone
Change from Baseline obesity incidence at 24 months | month 2, month 14 and month 24
  BMI value:
  * [25-30[ kg/m2 with a waist circumference above the norm (≥ 94cm for men or
    ≥ 80cm for women)
  * ≥ 30 kg/m2
Change from Baseline hypothyroidism incidence at 24 months | month 2, month 14 and month 24
  * level of thyroid-stimulating hormone
  * level of total thyroxine
Change from Baseline dyslipidemias incidence at 24 months | month 2, month 14 and month 24
  hypercholesterolemia (LDL) ≥ 1.6 g/L estimated by the Friedewald formula and/or a hypertriglyceridemia ≥ 4 g/L
Change from Baseline Heart failure markers incidence at 24 months | month 2, month 14 and month 24
  NT-proBNP and/or troponin I level above the threshold values.
Change from Baseline Atrial fibrillation incidence at 24 months | month 2, month 14 and month 24
  equivocal electrocardiogram, interpreted by an experienced physician
Change from Baseline of respiratory failure markers incidence at 24 months | month 2, month 14 and month 24
  FVC, FVC, FEV1, FEF25-75, FEF50, FEF25 (established by spirometric test) ≤ 80% of the predicted values (abacus on age, sex, height and origin ethnic)
Change from Baseline return to work issues incidence at 24 months | month 2, month 14 and month 24
  Diagnosed by a social worker
Change from Baseline of Lifestyle risk factors ( tobacco, alcohol, and cannabis) incidence at 24 months | month 2, month 4, month 14 and month 24
  consumption :
  * smoking and/or active cannabis
  * alcohols higher than the latest recommendations
Change from baseline Myelodysplastic syndromes and secondary acute leukemia incidence at 24 months | month 4, month 14 and month 24
  confirmed by the reference diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Mauricette MICHALLET, PhD, MD, Principal Investigator — Centre Leon Berard
Locations (1):
- Centre Léon Bérard, Lyon, France